CLINICAL TRIAL: NCT05340764
Title: Safety, Efficacy, and Cost-effectiveness of a Reduced Infliximab Infusion Time Protocol
Brief Title: Safety of Reduced Infliximab Infusion Time
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Chien-Huan Chen, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202007200
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2-hour infusion of infliximab (Active Comparator): 2 hour infusion of infliximab
  Infliximab: Infliximab is an effective and commonly used medication to treat patients with IBD. Patients in this group received the standard 2 hour infusion of infliximab and serves as the control group.
  Interventions: Drug: Infliximab
- 1-hour infusion of infliximab (Experimental): 1 hour infusion of infliximab
  Infliximab: Infliximab is an effective and commonly used medication to treat patients with IBD. Patients in this group received the reduced 1 hour infusion of infliximab and serves as the study group.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab is an effective and commonly used medication to treat patients with IBD

SUMMARY:
Remicade is a common medicine used for the treatment of inflammatory bowel disease. This medication is given as an intravenous infusion over 2 hours. Studies have suggested it is safe to give the infusion at a faster rate. The investigators would like to see if the infusion can be given over 1 hour. The investigators expect that increasing the rate of infusion WILL NOT lead to an increase in infusion reactions and will be just as safe and effective as the standard 2 hours dose.

DETAILED DESCRIPTION:
1.1 Infliximab use in IBD

Inflammatory bowel disease (IBD) affects 349 per 100,000 adults in the United States and is associated with significant morbidity and mortality. Infliximab is an effective and commonly used medication to treat patients with IBD, but a main safety concern is an antibody-induced infusion reaction. The incidence of infusion reactions is ~6.5%, with mild, moderate, or severe reactions occurring in 3.1%, 1.2%, and 1% of infusions, respectively. Because of the concern for infusions reactions, infliximab is FDA approved to be infused over 2 hours or more. The typical interval for infusions is every eight weeks but is at times reduced to every 4 weeks in patients with IBD. This infusion time represents a significant inconvenience to patients who receive regular maintenance infusions.

1.2 Accelerated Infliximab Infusions

Multiple studies outside of the United States have demonstrated that a shortened infusion time to one hour, and even thirty minutes is safe and tolerable with similar rates of infusion reactions compared to an infusion time of two hours. However, these studies have differed in dosing, interval, pre-medication allowed in the study, and they are not randomized controlled studies. It has also been shown that reducing infusion times leads to cost savings and increased patient satisfaction. A recent study conducted in the United States at the University of California in San Francisco, confirmed that a shortened infusion time of one hour is safe and tolerated.

1.3 Rationale

The hypothesis is that a shortened infusion time to one hour will be safe and tolerated, with equal infusion reaction rates compared to two-hour infusion

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age
2. Must have a diagnosis of IBD
3. Must be receiving Infliximab or biosimilar drug infusions for IBD at one of the study infusion centers - Center for Advanced Medicine, Barnes-Jewish West County, Barnes-Jewish South County infusion centers, or receiving infusion through BJC Home Care Services/ Barnes Home Health Company.
4. Must tolerate the three induction doses or be tolerating current maintenance dosing without an infusion reaction to qualify for randomization.

Exclusion Criteria:

1. Those receiving Infliximab for an indication other than IBD (the investigators will include patients receiving infliximab or biosimilar drug for both IBD and an additional autoimmune disease)
2. Patients with history of a moderate or severe infusion reactions to infliximab or to an infliximab biosimilar as defined in section 7
3. Patients with known antidrug antibodies to infliximab
4. Patients who are restarting infliximab (patients who have received infliximab within the past year but have now had an interval greater than 13 weeks between prior dose) must tolerate the three induction doses to qualify for randomization
5. Patients receiving an additional infusion concomitant with infliximab (e.g. IV iron)
6. Patients who decline to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abushamma S, Walker T, Garza K, Chen L, Nix D, Chen CH. Accelerated Infliximab Infusion Safety and Tolerability Is Non-inferior to Standard Infusion Protocol in Inflammatory Bowel Disease Patients: A Randomized Controlled Study. Crohns Colitis 360. 2023 May 3;5(3):otad022. doi: 10.1093/crocol/otad022. eCollection 2023 Jul. PMID 37288326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2020 to 2021 and followed throughout the study after enrollment. Patients aged 18 years or older with an established diagnosis of IBD, receiving infliximab at one of our infusions centers and have tolerated the 3 induction doses and current maintenance dosing were eligible for inclusion in the study.
Pre-assignment Details: Patients were excluded if they were receiving infliximab exclusively for a non-IBD indication, had a history of moderate or severe infusion reactions to infliximab (or biosimilar), had known antidrug antibodies to infliximab, had an interval greater than 13 weeks from prior dose of infliximab, were receiving an additional infusion concomitant with infliximab (eg, IV iron), or declined to participate in the trial.
Period: Overall Study
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Started | 45 | 51
Completed | 45 | 50
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1-hour Infusion of Infliximab: 1 hour infusion of infliximab
  Infliximab: Infliximab is an effective and commonly used medication to treat patients with IBD
- Total: Total of all reporting groups
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab | Total
Number analyzed (Participants) | 45 | 51 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age was 47 (SD 15.5) in both groups in the trial.
  years | 47 (15.5) | 47 (15.5) | 47 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 23 | 28 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 51 | 96
Inflammatory Bowel Disease Type [Count of Participants; unit: Participants]
  Ulcerative Colitis patients | 11 | 10 | 21
  Crohn's Disease patients | 34 | 41 | 75
Concomitant Immunomodulator [Count of Participants; unit: Participants]
  6-MP | 8 | 5 | 13
  AZA | 9 | 11 | 20
  MTX | 5 | 10 | 15
  None | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Infusion Reaction as Assessed by the Nursing Staff of the Infusion Unit
Description: Acute infusion reaction is defined as any reaction occurring during or within 1 hour after completion of the infusion. It will be separated into mild reactions and moderate/severe reactions as outlined below.
  Mild/Localized Reaction Pruritus Flushing (facial erythema) Rash/Urticaria Rigors Swelling Moderate/Severe Reaction Fever (temperature > 38.3 degree Celsius) Heart Rate greater than 120 Dyspnea/Shortness of breath Decrease in consciousness Hypotension defined as decrease in baseline SBP by >20 mmHg or SBP <85 Bronchospasm or laryngospasm Anaphylactic shock of one hour, to the standard two-hour infusion.
Time Frame: Median of 12 months in the control and a median of 14 months in the study group.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Number analyzed (Participants) | 45 | 51
Participants
  Mild Acute Infusion Reaction | 27 | 30
  Moderate/Severe Infusion Reaction | 0 | 0
  No Infusion Reaction | 18 | 21

2. Secondary Outcome: Cost Saving Analysis
Description: Direct costs of the 2 hour infusion per-infusion per-patient in dollar amount will be compared to direct costs of the 1 hour infusion per-infusion per-patient in dollar amount in our institution and the difference will be reported.
  Nursing Cost and Chair Occupancy Cost obtained from BJH Human Resources Department.
Time Frame: Median of 12 months in the control and a median of 14 months in the study group.
Measure: Mean (Full Range); unit: dollars
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Number analyzed (Participants) | 45 | 51
dollars
  Nursing Cost | 124.41 [106 to 413] | 72.57 [53 to 207]
  Chair Occupancy Cost | 350 [145 to 544] | 225 [72.50 to 272]

3. Secondary Outcome: Effect of Concomitant Immunomodulators and Pre-medications on Rate of Infusion Reactions - Median Number of Infusions
Description: Assess effect of concomitant immunomodulators and pre-medications on rate of infusion reactions - Median number of infusions
Time Frame: Median of 12 months in the control and a median of 14 months in the study group.
Measure: Median (Inter-Quartile Range); unit: Infusions
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Number analyzed (Participants) | 45 | 51
Infusions | 7 [5 to 8] | 7 [6 to 9]

4. Secondary Outcome: Number of Infusions Where Concomitant Immunomodulators and Pre-medications Were Used
Description: Number of Infusions where Concomitant Immunomodulators and Pre-medications were used in the study
Time Frame: Median of 12 months in the control and a median of 14 months in the study group.
Measure: Count of Units; unit: Total number of infusions
Units Other Than Participants: Total number of infusions
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Number analyzed (Participants) | 45 | 51
Number analyzed (Total number of infusions) | 309 | 376
Total number of infusions
  Premedications | 175 | 106
  Acetaminophen | 171 | 99
  Diphenhydramine | 110 | 69
  Loratidine | 7 | 11
  Ondansetron | 4 | 0
  Methylprednisolone | 4 | 1

5. Secondary Outcome: Effect of Concomitant Immunomodulators and Pre-medications on Rate of Infusion Reactions - Duration of Follow up (in Months)
Description: Assess effect of concomitant immunomodulators and pre-medications on rate of infusion reactions - Duration of follow up (in months)
Time Frame: Median of 12 months in the control and a median of 14 months in the study group.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
Number analyzed (Participants) | 45 | 51
months | 12 [8 to 16] | 14 [8 to 16]

ADVERSE EVENTS:
Time Frame: Up to 16 months
Arm/Group | 2-hour Infusion of Infliximab | 1-hour Infusion of Infliximab
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/51
Other Adverse Events (participants affected / at risk) | 0/45 | 0/51

LIMITATIONS AND CAVEATS:
1. We excluded pts. receiving induction doses of INX, pts. with a history of infusion reactions (IRR) and pts. with known antidrug antibodies to INX, as studies have shown an increased infusion reaction rate in these pts. This may have contributed to the absence of clinically significant infusion reactions.
2. We did not assess delayed IRR, as they occur at a much lower rate than acute IRR.
3. Majority of pts. assessed for eligibility were excluded primarily due to various reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT05340764/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05340764/ICF_001.pdf